CLINICAL TRIAL: NCT01206309
Title: Longitudinal Study of Immune Mediated Disorders After Allogeneic Hematopoietic Cell Transplantation (HCT)
Brief Title: Immune Mediated Disorders After Allogeneic Hematopoietic Cell Transplantation
Status: Completed | Type: Observational
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: RDCRN 6501; U54CA163438 (NIH); RDCRN-6501 (Other: DMCC); 2342.00 (Other: FHCRC)
Record Dates: First submitted 2010-09-20; First posted 2010-09-21 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Graft vs Host Disease; Cutaneous Sclerosis; Bronchiolitis Obliterans
Keywords: Graft vs Host Disease; Allogeneic Hematopoietic Cell Transplantation; Bone Marrow Transplantation; Peripheral Blood Stem Cell Transplantation; Umbilical Cord Blood Stem Cell Transplantation
MeSH Terms: conditions — Graft vs Host Disease; Bronchiolitis Obliterans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and urine specimens
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Controls: Never develop an immune mediated disorder
- Immune Mediated Disorder: Develop an immune mediated disorder

SUMMARY:
The purpose of this research study is to better understand the onset and course of graft versus host disease (GVHD)and other immune-mediated disorders after stem cell transplant.

DETAILED DESCRIPTION:
Allogeneic hematopoietic cell transplantation (HCT) is the only known curative option for many hematologic disorders. After transplantation, many patients develop immune mediated disorders that may be life-threatening such as graft versus host disease (GVHD). The morbidity and mortality associated with HCT-associated immune mediated disorders are major barriers to successful use of transplantation to cure rare hematologic malignancies such as leukemia, lymphoma, multiple myeloma, myelodysplastic/myeloproliferative syndromes amongst other diseases.

With this study, the investigators will investigate the biologic basis for immune mediated disorders after allogeneic HCT, focusing on those developing cutaneous sclerosis, bronchiolitis obliterans syndrome, late acute GVHD and chronic GVHD. The study will enroll 1118 (1018 adults and 100 children) allogeneic HCT patients over a three year period. Subjects will be followed for two years and monitored closely for development of immune mediated disorders. This study will have 5 study visits at day 1, 100, 180, 365, and 730. During these visits, a physical assessment, medication review, blood and urine collection will occur.

If a subject develops an immune mediated disordered, they will be monitored at 3 months, 6 months, 1 year and then annually from the date of diagnosis. During these study visits, a physical assessment, IMD status, and medication review as well as blood and urine collection will occur.

ELIGIBILITY:
Inclusion Criteria:

* Planned or completed first allogeneic stem cell transplant (any conditioning regimen, graft source, donor type and GVHD prophylaxis regimen)
* Signed, informed consent and, if applicable, child assent

Exclusion Criteria:

* Inability to comply with study procedures
* Anticipated survival less than 6 months due to co-morbid disease
* Autoimmune disorder or inherited immunodeficiency before HCT
* Diagnosis of late acute or chronic GVHD prior to study enrollment
* Hematologic relapse or chemotherapy refractory disease at restaging within 1 month of HCT or at the time of enrollment (e.g., > 5% blasts for leukemia; poorly responsive lymphoma)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are preparing for or have recently received an allogeneic hematopoietic cell transplant
Sampling Method: Probability Sample
Enrollment: 911 (Actual)
Dates: Start 2011-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
The prevalence of immune mediated disorders | Diagnosis of IMD and at 2 years
  The prevalence of:
  * Persistent, recurrent or late onset acute GVHD
  * Cutaneous Sclerosis
  * Bronchiolitis Obliterans Syndrome
  * Chronic GVHD

SECONDARY OUTCOMES:
Banked blood and urine samples | At 2 years
  Summarized as the percentage of compliance for each center and for the study as a whole

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Lee, MD, MPH, Principal Investigator — Fred Hutchinson Cancer Center
Locations (14):
- United States (14):
  - Mayo Clinic, Scottsdale, Arizona
  - Stanford University, Stanford, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University St. Louis, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Cornell Medical College, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Vanderbilt University, Nashville, Tennessee
  - Fred Hutchinson Cancer Research Center/Seattle Cancer Care Alliance, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Filipovich AH, Weisdorf D, Pavletic S, Socie G, Wingard JR, Lee SJ, Martin P, Chien J, Przepiorka D, Couriel D, Cowen EW, Dinndorf P, Farrell A, Hartzman R, Henslee-Downey J, Jacobsohn D, McDonald G, Mittleman B, Rizzo JD, Robinson M, Schubert M, Schultz K, Shulman H, Turner M, Vogelsang G, Flowers ME. National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease: I. Diagnosis and staging working group report. Biol Blood Marrow Transplant. 2005 Dec;11(12):945-56. doi: 10.1016/j.bbmt.2005.09.004. PMID 16338616